CLINICAL TRIAL: NCT04263584
Title: A Prospective Multicenter Phase 2 Study of Copanlisib in Combination With Rituximab and CHOP Chemotherapy (COPA-R-CHOP) in Patients With Previously Untreated Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Copanlisib in Combination With Rituximab and CHOP Chemotherapy in Patients With Previously Untreated DLBCL
Acronym: COPA-R-CHOP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM18-0021
Record Dates: First submitted 2020-01-07; First posted 2020-02-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Copanlisib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — copanlisib; R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Copanlisib and R-CHOP chemotherapy (Experimental): All patients will receive 6 cycles of R-CHOP immunochemotherapy every two weeks with the following doses per cycle: rituximab 375 mg/m², cyclophosphamide 750 mg/m², doxorubicin 50 mg/ m², vincristine 1.4 mg/m² (dose capped at 2 mg or 1 mg for individuals above 60 years of age), prednisolone 500 mg. In addition, copanlisib at a dose of 60 mg will be administered on days 1 and 8 of each 21-day cycle of R-CHOP in the first 6 patients. If dose limiting toxicity (DLT) occurs in no more than one out of these 6 patients during cycle 1, additional 6 patients at 60 mg will be enrolled and treated for at least 1 cycle before opening the phase II portion of the study. If a DLT is observed in 2 or more of the first 6 patients during cycle 1 the dose of copanlisib will be reduced to 45 mg on days 1 and 8 for the next 6 patients. The data of the safety run-in analysis (first 12 patients) will be presented to the Data Safety Monitoring Board and the recommended phase 2 dose will be determined.
  Interventions: Drug: Copanlisib; Drug: R-CHOP Chemotherapy

INTERVENTIONS:
Drug: Copanlisib — Copanlisib vials 60 mg
Drug: R-CHOP Chemotherapy — Immunochemotherapy

SUMMARY:
This is a prospective, multicenter, non-randomized, open-label, phase II study to describe the efficacy of R-CHOP plus copanlisib including a safety run-in phase in order to detect early and common unexpected toxicities caused by the addition of copanlisib to the standard immuno-chemotherapy R-CHOP in patients with diffuse large B-cell lymphoma (DLBCL)

DETAILED DESCRIPTION:
Patients diagnosed with DLBCL can be cured with a combined approach of CHOP chemotherapy and the anti-CD20 antibody rituximab in roughly 65% of cases. About one third of patients with DLBCL relapse or show primary progressive disease after modern first-line therapy. The outcome of these patients is poor in particular if first-line therapy contained rituximab. Novel therapeutic approaches are urgently warranted. Thus, it is the goal to further improve progression-free Survival (PFS) and overall Survival (OS) by combining R-CHOP with copanlisib. Copanlisib is a small molecule pan-class 1 PI3K inhibitor and approved by US FDA for the treatment of adult patients with relapsed follicular lymphoma who have received at least two prior systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed

   1. DLBCL (NOS) or
   2. High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements or
   3. High-grade B-cell lymphoma (NOS)
   4. Follicular lymphoma Grade 3B (primary diagnosis without history of indolent lymphoma) with a diagnostic biopsy performed within 3 months before study entry and with material available for central review and complimentary scientific analyses
2. 18-80 years of age
3. International Prognostic Index (IPI) 2-5
4. Eastern Cooperative Oncology Group Performance status (ECOG) 0-2
5. Life expectancy of at least 3 months
6. Women of childbearing potential and men must agree to use effective contraception when sexually active. This applies for the time period between signing of the informed consent form and 6 months after the last administration of study treatment. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control (failure rate of less than 1%), e.g. intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner and sexual abstinence. The use of condoms by male patients is required unless the female partner is permanently sterile.

   Adequate baseline laboratory values collected no more than 7 days before starting study treatment:
7. Total bilirubin ≤ 1.5 x ULN (< 3 x ULN for patients with Gilbert syndrome, patients with cholestasis due to compressive adenopathies of the hepatic hilum or documented liver involvement or with biliary obstruction due to lymphoma)
8. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement by lymphoma)
9. Lipase ≤ 1.5 x ULN
10. Glomerular filtration rate (GFR) ≥ 40 mL/min/1.73 m2 according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. If not on target, this evaluation may be repeated once after at least 24 hours either according to the CKD-EPI formula or by 24-hour sampling. If the later result is within acceptable range, it may be used to fulfill the inclusion criteria instead.
11. INR and PTT ≤ 1.5 x ULN
12. Platelet count ≥ 75,000 /mm3.
13. Hemoglobin (Hb) ≥ 8 g/dL
14. Absolute neutrophil count (ANC) ≥ 1,500/mm3
15. Left ventricular ejection fraction ≥ 50%
16. No prior lymphoma therapy
17. Ability to understand and willingness to sign written informed consent. Signed informed consent must be obtained before any study specific procedure.

Exclusion Criteria:

Patients who meet any of the following criteria at the time of screening will be excluded.

1. Previous assignment to treatment during this study. Patients permanently withdrawn from study participation will not be allowed to re-enter the study.
2. Previous (within 28 days or less than 5 half-lives of the drug before start of study treatment) or concomitant participation in another clinical study with investigational medicinal product(s).
3. Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent persons (e.g. employee or student of the investigational site).

   Excluded medical conditions:
4. Type I or II diabetes mellitus with HbA1c > 8.5% at screening or fasting plasma glucose > 160 mg/dL at screening
5. History or concurrent condition of interstitial lung disease and/or severely impaired lung function (as judged by the investigator)
6. Known lymphoma involvement of the central nervous system
7. Human immunodeficiency virus (HIV) infection
8. Hepatitis B (HBV) and C (HCV) infection. Patients with serologic markers of HBV immunization due to vaccination (HBsAg negative, Anti-HBc negative and Anti-HBs positive) will be eligible
9. CMV-PCR positive at baseline
10. Previous or concurrent history of malignancies within 5 years prior to study treatment except for curatively treated:

    1. Cervical carcinoma in situ
    2. Non-melanoma skin cancer
    3. Superficial bladder cancer (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria])
    4. Localized prostate cancer
11. Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication
12. Patients with seizure disorder requiring medication
13. Proteinuria of ≥ CTCAE Grade 3 as assessed by a 24h protein quantification or estimated by urine protein: creatinine ratio > 3.5 on a random urine sample
14. Concurrent diagnosis of pheochromocytoma
15. Congestive heart failure > New York Heart Association (NYHA) class 2
16. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
17. Myocardial infarction less than 6 months before start of test drug
18. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
19. Non-healing wound, ulcer, or bone fracture
20. Active, clinically serious infections > CTCAE Grade 2
21. Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management)
22. Known history of drug induced liver injury, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, on-going extra-hepatic obstruction caused by cholelithiasis, cirrhosis of the liver or portal hypertension
23. Ongoing inflammatory bowel disease
24. History of, or current autoimmune disease
25. Prior treatment with PI3K inhibitors
26. Any other co-existing medical or psychological condition that will preclude participation in the study or compromise ability to give informed consent
27. Patient is pregnant (β-HCG positive) or breast-feeding
28. Known hypersensitivity to copanlisib or to any of the excipients of rituximab, cyclophosphamide, doxorubicine, vincristine, and/or prednisone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | From the day of inclusion into the study until event (disease progression, relapse, death due to any other cause) occurs, assessed up to 4 years.
  Length of time that a patient lives without disease progression or relapse.

SECONDARY OUTCOMES:
Overall survival | From the day of inclusion into the study to death due to any cause, assessed up to 4 years.
  The percentage of patients in this study who are still alive.
Event-free survival | From the day of inclusion into the study until event (disease progression, start of additional, unplanned anti-tumor therapy, relapse, death due to any other cause) occurs, assessed up to 4 years.
  Length of time that a patient remains free of certain events (disease progression, start of additional, unplanned antitumor therapy, relapse, death due to any other cause).
Rate of complete remission | From the day of inclusion into the study until date of complete remission, assessed up to 4 years.
  Rate of complete remission measured as number of complete remissions divided by the number of patients included.
Rate of partial remission | From the day of inclusion into the study until date of partial remission, assessed up to 4 years.
  Rate of partial remission measured as number of partial remissions divided by the number of patients included.
Overall response rate | From the day of inclusion into the study until date of complete or partial remission, assessed up to 4 years.
  Overall response rate measured as number of complete and partial remissions divided by the number of patients included.
Progression rate | From the day of inclusion into the study until date of progression during therapy or within 2 months after last treatment course.
  Progression rate measured as number of progressions divided by the number of patients included.
Relapse rate | From the day of inclusion into the study until date of relapse during therapy or within 2 months after last treatment course.
  Relapse rate measured as number of relapses divided by the number of patients included.
Duration of response | From documentation of tumor response to relapse, assessed up to 4 years.
  The time between the initial response to therapy and subsequent disease progression or relapse.
Adverse events and serious adverse events | The documentation of adverse events, including serious adverse events, starts with first study treatment after patient inclusion and ends 100 days after the last application of copanlisib or any component of R-CHOP
  Frequency of adverse events and serious adverse events
Rate of treatment-related deaths | From the start of therapy up to 2 months after the end of therapy.
  The number of deaths during therapy or up to 2 months after the end of therapy divided by the number of patients included.
Therapy cycles (number) | From the start of therapy (copanlisib and R-CHOP) until the end of therapy (last application of copanlisib or any component of R-CHOP), assessed up to 0.5 years.
  Number of therapy cycles
Therapy cycles (duration) | From the start of therapy (copanlisib and R-CHOP) until the end of therapy (last application of copanlisib or any component of R-CHOP), assessed up to 0.5 years.
  Duration of therapy cycles
Used drugs | From the start of therapy (copanlisib and R-CHOP) until the end of therapy (last application of copanlisib or any component of R-CHOP), assessed up to 0.5 years.
  Cumulative doses of R-CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone, rituximab) and copanlisib.
Outcome according to lymphoma biology | From the start of study until the end of study, assessed up to 4 years.
  Lymphoma tissue from all patients will be characterized.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Georg Lenz, MD, Principal Investigator — University Hospital Muenster
Locations (12):
- Germany (12):
  - University Hospital RWTH Aachen, Aachen
  - Klinikum-Bremen-Mitte, Bremen
  - St.-Johannes-Hospital Dortmund, Dortmund
  - Onkozentrum Dresden, Dresden
  - University Hospital Halle, Halle
  - Westpfalz-Klinikum, Kaiserslautern
  - ÜBAG MVZ Dr. Vehling-Kaiser GmbH, Landshut
  - University Hospital Leipzig, Leipzig
  - Hospital of the Ludwig-Maximilians-University (LMU) Munich, Munich
  - University Hospital Muenster, Münster
  - Hospital Stuttgart - Stuttgart Cancer Center, Stuttgart
  - University Hospital Ulm, Ulm